CLINICAL TRIAL: NCT02535611
Title: Evaluation of Memantine Versus Placebo on Ischemic Stroke Outcome
Acronym: EMISO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mazandaran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Nasim Tabrizi, Assistant professor of neurology, Mazandaran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MAZUMS
Record Dates: First submitted 2015-08-22; First posted 2015-08-28 (Estimated); Results first posted 2020-09-16 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-09

CONDITIONS: Ischemic Stroke; Excitotoxicity; Memantine
MeSH Terms: conditions — Ischemic Stroke | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Memantine (Active Comparator): Patients with ischemic stroke in middle cerebral artery (MCA) territory who will receive 20 mg/d(2 tab 5mg BID) memantine for 7 days and then 10mg/d(1 tab 5mg BID) memantine for 21 days.
  Interventions: Drug: Memantine
- Placebo (Placebo Comparator): Patients with ischemic stroke in middle cerebral artery (MCA) territory who will receive placebo(2 tab BID) for 7 days and continue placebo(1 tab BID) for 21 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Beside the usual treatment of ischemic stroke, this group will receive placebo for 4 weeks.
  Arms: Placebo
Drug: Memantine — Beside the usual treatment for ischemic stroke this group will be treated by memantine.
  Arms: Memantine

SUMMARY:
The researchers aim to investigate the effect of memantine on stroke outcome in a randomized double-blind placebo-controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Presentation at first 24hrs of disease onset
* Confirmation of ischemic stroke in MCA territory by imaging.
* Accepted consent form

Exclusion Criteria:

* Allergy history to memantine
* Stage 4 -5 renal failure base on Acute Kidney Injury Network criteria
* Moderate to severe hepatic failure (Child-Pugh criteria, grade B and C)
* History of epilepsy
* History of dementia
* History of memantine use in recent 6 months
* Pregnancy or breastfeeding
* Severe drug adverse effects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-09 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Memantine | Placebo
Started | 27 | 20
Completed | 27 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Memantine | Placebo | Total
Number analyzed (Participants) | 27 | 20 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 8 | 18
  >=65 years | 17 | 12 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.56 (13.03) | 69.75 (14.61) | 70.79 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 7 | 21
  Male | 13 | 13 | 26
Region of Enrollment [Number; unit: participants]
  Iran | 27 | 20 | 47

OUTCOME MEASURES:

1. Primary Outcome: Investigation of Neurological Deficit by National Institute of Health Scale Score (NIHSS)
Description: The National Institutes of Health Stroke Scale, or NIH Stroke Scale (NIHSS) is a tool used by healthcare providers to objectively quantify the impairment caused by a stroke. The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment. The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0. Higher score is indicative of some level of impairment in neurological function.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 27 | 20
score on a scale | 4.52 (4.51) | 5.75 (4.94)

2. Primary Outcome: Investigation of Disability by Modified Rankin Scale (mRS)
Description: The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability.
  The scale runs from 0-6, running from perfect health without symptoms to death.
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 27 | 20
score on a scale | 2.89 (0.75) | 2.55 (1.19)

3. Secondary Outcome: Investigation of Neurological Deficit by National Institute of Health Scale Score (NIHSS)
Description: as for outcome 1
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 27 | 20
score on a scale | 3.42 (2.96) | 4.4 (3.98)

4. Secondary Outcome: Investigation of Disability by Modified Rankin Scale (mRS)
Description: as for outcome 2
Time Frame: 28 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 27 | 20
score on a scale | 2.3 (0.95) | 2.3 (1.3)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Memantine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/20
Other Adverse Events (participants affected / at risk) | 0/27 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes